CLINICAL TRIAL: NCT03260205
Title: A Phase 3, Randomized, Double-blind, Multicenter, Parallel-group, Placebo-controlled, Fixed-Dose Safety and Efficacy Study of SPD489 Compared With Placebo in Preschool Children Aged 4-5 Years With Attention-deficit/Hyperactivity Disorder
Brief Title: Safety and Efficacy Study in Preschool Children Aged 4-5 Years With Attention-deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPD489-347
Record Dates: First submitted 2017-08-09; First posted 2017-08-24 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: SPD489; Lisdexamfetamine dimesylate; ADHD; hyperactivity; Neurobehavioral disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participant will receive placebo matching to SPD489 (Lisdexamfetamine dimesylate) capsule for 6 weeks.
  Interventions: Drug: Placebo
- SPD489 (Lisdexamfetamine dimesylate) (Experimental): Participants will be randomized to receive SPD489 capsule in a 5:5:5:5:6 ratio to SPD489 5, 10, 20, 30 milligram (mg) orally once daily for 6 weeks. Dosing will begin with the lowest strength of SPD489 (5 mg), and will be titrated until the randomly assigned fixed-dose is reached.
  Interventions: Drug: SPD489 (Lisdexamfetamine dimesylate); Drug: SPD489

INTERVENTIONS:
Drug: Placebo — Placebo matching to SPD489 (Lisdexamfetamine dimesylate) capsule for 6 weeks.
  Arms: Placebo
Drug: SPD489 (Lisdexamfetamine dimesylate) — SPD489 capsule in a 5:5:5:5:6 ratio to 5, 10, 20, 30 mg orally once daily for 6 weeks.
  Arms: SPD489 (Lisdexamfetamine dimesylate)
Drug: SPD489 — SPD489
  Arms: SPD489 (Lisdexamfetamine dimesylate)

SUMMARY:
The purpose of this study is to determine if an investigational treatment is effective in improving the total score on the ADHD-RS-IV Preschool Version in children 4-5 years old diagnosed with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a male or female aged 4-5 years inclusive at the time of consent
* Participant's parent(s) or legally authorized representative (LAR) must provide signature of informed consent, and there must be documentation of assent (if applicable) by the participant before completing any study related procedures.
* Participant and parent(s)/LAR are willing and able to comply with all of the testing and requirements defined in the protocol, including oversight of morning dosing.
* Participant must meet DSM-IV-TR criteria for a primary diagnosis of ADHD (any sub-type).
* Participant has an ADHD-RS-IV Preschool Version Total Score at the baseline visit (Visit 0) greater than or equal to 28 for boys, and greater than or equal to 24 for girls.
* Participant has a Clinical Global Impressions - Severity of Illness (CGI-S) score greater than or equal to 4 at the baseline visit (Visit 0).
* Participant has a Peabody Picture Vocabulary Test standard score of greater than or equal to 70 at the screening visit (Visit -1).
* Participant has undergone an adequate course of non-pharmacological treatment or has a severe enough condition to consider enrollment without undergoing prior non-pharmacological treatment.
* Participant has participated in a structured group activity (e.g, preschool, sports, Sunday school) so as to assess symptoms and impairment in a setting outside the home.
* Participant has lived with the same parent(s) or guardian for greater than or equal to 6 months.

Exclusion Criteria:

* Participant is required to or anticipates the need to take any prohibited medications or medications that have central nervous system (CNS) effects or have an effect on performance. Stable use of bronchodilator inhalers is not exclusionary.
* Participant has taken another investigational product or has taken part in a clinical study within 30 days prior to the screening visit (Visit -1).
* Participant is well-controlled on his/her current ADHD medication with acceptable tolerability.
* Participant has a concurrent chronic or acute illness, disability, or other condition that might confound the results of safety assessments or may increase risk to the participant..
* Participant has glaucoma.
* Participant has failed to fully respond to an adequate course of amphetamine therapy.
* Participant has a documented allergy, hypersensitivity, or intolerance to amphetamine or to any excipients in the investigational product.
* Participant has a known family history of sudden cardiac death or ventricular arrhythmia.
* Participant has a blood pressure measurement greater than or equal to 95th percentile for age, sex, and height at the screening visit (Visit -1) or the baseline visit (Visit 0) or history of moderate or severe hypertension.
* Participant has a known history of symptomatic cardiovascular disease, unexplained syncope, exertional chest pain,advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems.
* Participant has any clinically significant clinical laboratory abnormalities at the screening visit (Visit -1) or electrocardiogram (ECG) at screening visit (Visit-1) or baseline visit (Visit 0) based on investigator judgment.
* Participant has current abnormal thyroid function, defined as abnormal thyroid stimulating hormone (TSH) and thyroxine (T4) at the screening visit (Visit -1). Treatment with a stable dose of thyroid medication for at least 3 months is permitted.
* Participant has a current, controlled (requiring medication or therapy) or uncontrolled, co-morbid psychiatric disorder including but not limited to any of the below co-morbid Axis I disorders and Axis II disorders:

  i. post-traumatic stress disorder or adjustment disorder ii. bipolar illness, psychosis, or a family history of these disorders iii. pervasive developmental disorder iv. obsessive-compulsive disorder (OCD) v. psychosis/schizophrenia vi. a serious tic disorder, or a family history of Tourette's disorder vii. Participant is currently considered a suicide risk in the opinion of the investigator, has previously made a suicide attempt, or has a prior history of, or is currently demonstrating active suicidal ideation.

viii. a history of physical, sexual, or emotional abuse ix. any other disorder or agitated state that in the opinion of the investigator, contraindicates SPD489 or lisdexamfetamine dimesylate treatment or confound efficacy or safety assessments.

* Participant has initiated behavioral therapy within 1 month of the baseline visit (Visit 0). Participant may not initiate behavioral therapy during the study.
* Participant has a height less than equal to (<=) 5th percentile for age and sex at the screening visit (Visit -1).
* Participant has a weight <= 5th percentile for age and sex at the screening visit (Visit -1).
* Participant lives with anyone who currently abuses stimulants or cocaine.
* Participant has a history of seizures (other than infantile febrile seizures).
* Participant is taking any medication that is excluded per the protocol.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 199 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (48):
- United States (48):
  - Harmonex, Inc, Dothan, Alabama
  - Preferred Research Partners, Inc, Little Rock, Arkansas
  - CMB Clinical Trials, Colton, California
  - Sun Valley Research Center, Imperial, California
  - Alliance for Wellness d/b/a Alliance for Research, Long Beach, California
  - Asclepes Research, Panorama City, California
  - Psychiatric Centers at San Diego, San Diego, California
  - UCSF Dept of Psychiatry, San Francisco, California
  - Elite Clinical Trials, Inc, Wildomar, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - APG Research, LLC, Orlando, Florida
  - University of South Florida, St. Petersburg, Florida
  - University of South Florida Department Of Psychiatry, Tampa, Florida
  - iResearch Atlanta LLC, Decatur, Georgia
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Clinical Neurophysiology Services, Sterling Heights, Michigan
  - Washington University, St Louis, Missouri
  - Premier Psychiatric Reseach Institute, LLC, Lincoln, Nebraska
  - Jersey Shore University Medical Center (JSUMC), Neptune City, New Jersey
  - Manhattan Behavioral Medicine, New York, New York
  - University of Rochester, Rochester, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Pediatric Associates of Fairfield, Inc, Fairfield, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Cyn3rgy Research Center, Gresham, Oregon
  - Rainbow Research Inc, Barnwell, South Carolina
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - Coastal Carolina Research, Mt. Pleasant, South Carolina
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - BioBehavioral Research of Austin, Austin, Texas
  - Bayou City Research Limited, Houston, Texas
  - BI Research Center, Houston, Texas
  - Red Oak Psychiatry Associates, Houston, Texas
  - Road Runner Research, San Antonio, Texas
  - Family Psychiatry of the Woodlands, The Woodlands, Texas
  - Ericksen Research and Development, Clinton, Utah
  - Clinical Research Partners, LLC, Petersburg, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Seattle Childrens Hospital, Pearl Clinic, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Childress AC, Lloyd E, Jacobsen L, Gunawardhana L, Johnson SA Jr, Findling RL. Efficacy and Safety of Lisdexamfetamine in Preschool Children With Attention-Deficit/Hyperactivity Disorder. J Am Acad Child Adolesc Psychiatry. 2022 Dec;61(12):1423-1434. doi: 10.1016/j.jaac.2022.03.034. Epub 2022 May 13. PMID 35577034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 49 sites in United States between 06 September 2017 (first participant enrolled) and 23 October 2018 (last participant completed).
Pre-assignment Details: A total of 284 participants were screened of them 85 participants were screen failures and did not receive any treatment. 199 participants (153 participants for SPD489 treatment and 46 participants for placebo treatment) were randomized, out of them 150 participants completed the study.
Groups:
- Placebo: Participants received placebo matched to SPD489 capsule orally once daily for 6 weeks.
- SPD489 5 mg: Participants received SPD489 5 mg capsule orally once daily for 6 weeks.
- SPD489 10 mg: Participants received SPD489 10 mg capsule orally once daily for 6 weeks.
- SPD489 20 mg: Participants received SPD489 20 mg capsule orally once daily for 6 weeks.
- SPD489 30 mg: Participants received SPD489 30 mg capsule orally once daily for 6 weeks.
Period: Overall Study
Arm/Group | Placebo | SPD489 5 mg | SPD489 10 mg | SPD489 20 mg | SPD489 30 mg
Started | 46 | 40 | 37 | 37 | 39
Received Treatment | 45 | 39 | 35 | 34 | 38
Completed | 37 | 32 | 26 | 30 | 25
Not Completed | 9 | 8 | 11 | 7 | 14
Not completed — Adverse Event | 2 | 0 | 2 | 2 | 4
Not completed — Lost to Follow-up | 2 | 2 | 1 | 1 | 5
Not completed — Protocol Violation | 0 | 0 | 2 | 0 | 1
Not completed — Withdrawal by Participant or Parent/LAR | 4 | 5 | 1 | 0 | 2
Not completed — Other: Unspecified | 0 | 0 | 3 | 1 | 1
Not completed — Participant Who Did Not Received AnyDose | 1 | 1 | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisted of all randomized set who had taken at least 1 dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SPD489 5 mg | SPD489 10 mg | SPD489 20 mg | SPD489 30 mg | Total
Number analyzed (Participants) | 45 | 39 | 35 | 34 | 38 | 191
Age, Continuous [Mean (Standard Deviation); unit: months] | 61.9 (6.32) | 60.7 (6.32) | 60.9 (7.18) | 61.1 (5.88) | 61.2 (7.23) | 61.2 (6.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 13 | 10 | 11 | 62
  Male | 29 | 27 | 22 | 24 | 27 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 11 | 2 | 5 | 32
  Not Hispanic or Latino | 37 | 33 | 24 | 32 | 33 | 159
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 19 | 17 | 18 | 18 | 17 | 89
  Race: Black or African American | 23 | 20 | 15 | 15 | 16 | 89
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Race: Multiple | 1 | 1 | 0 | 1 | 3 | 6
  Race: Other: Not specified | 1 | 1 | 2 | 0 | 1 | 5
  Race: Missing | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinician-Administered Attention-Deficit/Hyperactivity Disorder Rating Scale-IV (ADHD-RS-IV) Preschool Version Total Score at Week 6
Description: ADHD-RS-IV Preschool Version was adapted from the ADHD Rating Scale-IV and provided examples appropriate for the developmental level of preschool children. The ADHD-RS-IV Preschool Version was an 18-item questionnaire that required the respondent to rate the frequency of occurrence of ADHD symptoms as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition-Text Revision (DSM-IV-TR) criteria. Each item was scored on a 4-point scale ranging from 0 (never or rarely) to 3 (very often) with total scores ranging from 0-54. The 18 items were grouped into 2 subscales: hyperactivity/impulsivity (even numbered items 2-18) and inattentiveness (odd numbered items 1-17). Full analysis set (FAS) consisted of all participants in the safety analysis set who had at least 1 post-dose ADHD RS IV preschool version total score assessment.
Time Frame: Baseline, Week 6
Population: Full analysis set. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure. This outcome was pre-specified to collect and analyze pooled groups of SPD489 doses. The data were planned, analyzed, and reported only for the placebo and the pooled 10, 20, 30 mg doses of SPD489 arms.
Measure: Mean (Standard Error); unit: Score on a scale
Groups:
- Pooled SPD489 Doses (10, 20, and 30 mg): Participants received SPD489 10, 20, and 30 mg capsule orally once daily for 6 weeks were pooled.
Arm/Group | Placebo | Pooled SPD489 Doses (10, 20, and 30 mg)
Number analyzed (Participants) | 37 | 84
Score on a scale | -9.1 (2.36) | -14.2 (1.57)
Statistical Analysis 1: Comparison: Placebo vs Pooled SPD489 Doses (10, 20, and 30 mg); This outcome measure was analyzed using the linear mixed-effects model for repeated measures (MMRM). From a MMRM analysis over all post-baseline visits, with the change from baseline in ADHD-RS-IV preschool version total score as the outcome, treatment, visit, and treatment-by-visit interaction as fixed effect, baseline ADHD-RS-IV and baseline ADHD-RS-IV score-by-visit interaction as covariates; Test type: Superiority; p = 0.0242, MMRM; Difference in Least Square Mean = -5.9, 95% CI 2-sided [-11.01 to -0.78]

2. Secondary Outcome: Clinical Global Impressions Global Improvement (CGI-I) at Week 6
Description: CGI-I was an overall assessment of global symptom improvement by evaluation of the participant's condition severity and improvement over time. Scoring was done based on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse), where higher score reported worse condition. The scoring was elaborated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse. FAS consisted of all participants in the safety analysis set who had at least 1 post-dose ADHD RS IV preschool version total score assessment.
Time Frame: Week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Pooled SPD489 Doses (10, 20, and 30 mg)
Number analyzed (Participants) | 37 | 84
Score on a scale | 3.4 (0.18) | 2.8 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Pooled SPD489 Doses (10, 20, and 30 mg); This outcome measure was analyzed using the linear mixed-effects model for repeated measures (MMRM). From a MMRM analysis over all post-baseline Visits, with the CGI-I score as the outcome, treatment, visit, and treatment-by-visit interaction as fixed effect, baseline CGI-S as covariate; Test type: Superiority; p = 0.0074, MMRM; Difference in Least Mean Square = -0.6, 95% CI 2-sided [-1.03 to -0.16]

3. Secondary Outcome: Dose Response Relationship for Change From Baseline in ADHD-RS-IV Preschool Version Total Score in Preschool Children at Week 6
Description: Dose response relationship was evaluated by using the ADHD-RS Preschool Version Total Score. ADHD-RS-IV Preschool Version was adapted from the ADHD Rating Scale-IV and provided examples appropriate for the developmental level of preschool children. The ADHD-RS-IV Preschool Version was an 18-item questionnaire that requires the respondent to rate the frequency of occurrence of ADHD symptoms as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition-Text Revision (DSM-IV-TR) criteria. Each item was scored on a 4-point scale ranging from 0 (never or rarely) to 3 (very often) with total scores ranging from 0-54. The 18 items were grouped into 2 subscales: hyperactivity/impulsivity (even numbered items 2-18) and inattentiveness (odd numbered items 1-17). Dose response analysis set consisted of all participants in the safety analysis set who had at least 1 valid primary efficacy measurement on the randomized target dose level of the investigational product.
Time Frame: Baseline, Week 6
Population: Dose response analysis set. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure. Each SPD489 arm is compared with placebo sequentially, with the highest dose level first.
Measure: Mean (Standard Error); unit: Score on a scale
Groups:
- SPD489 30 mg: Participants received fixed dose of SPD489 30 mg capsule orally once daily for 6 weeks.
- SPD489 20 mg: Participants received fixed dose of SPD489 20 mg capsule orally once daily for 6 weeks.
- SPD489 10 mg: Participants received fixed dose of SPD489 10 mg capsule orally once daily for 6 weeks.
- SPD489 5 mg: Participants received fixed dose of SPD489 5 mg capsule orally once daily for 6 weeks.
Arm/Group | Placebo | SPD489 30 mg | SPD489 20 mg | SPD489 10 mg | SPD489 5 mg
Number analyzed (Participants) | 37 | 26 | 30 | 26 | 33
Score on a scale | -9.1 (2.36) | -15.3 (2.62) | -17.0 (2.90) | -10.8 (2.63) | -13.5 (2.53)

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a investigational product (IP) and that does not necessarily had a causal relationship with this treatment. TEAEs were defined as AEs that start or deteriorate on or after the date of the first dose of IP and no later than 3 days following the last dose of IP.
Time Frame: From start of study drug administration up to follow-up (Week 7)
Population: Safety analysis set consisted of all randomized set who had taken at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SPD489 5 mg | SPD489 10 mg | SPD489 20 mg | SPD489 30 mg
Number analyzed (Participants) | 45 | 39 | 35 | 34 | 38
Participants | 19 | 13 | 15 | 18 | 22

5. Secondary Outcome: Number of Participants With Potentially Clinically Significant Changes in Vital Signs
Description: Vital sign assessments included blood pressure (systolic and diastolic), average pulse rate. Number of participants with potentially clinically significant changes in vital signs were reported. mmHg represents millimetre of mercury in the outcome measure data.
Time Frame: Week 6
Population: Safety analysis set consisted of all randomized set who had taken at least 1 dose of investigational product. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SPD489 5 mg | SPD489 10 mg | SPD489 20 mg | SPD489 30 mg
Number analyzed (Participants) | 41 | 34 | 32 | 33 | 32
Participants
  Pulse: >=130 beats per minute (bpm), Week 6 | 0 | 0 | 0 | 0 | 0
  Pulse: <=55 bpm, Week 6 | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure (BP): >=120 mmHg, Week 6 | 0 | 0 | 0 | 1 | 0
  Systolic BP: <75 mmHg, Week 6 | 0 | 0 | 0 | 0 | 0
  Diastolic BP: >=85 mmHg, Week 6 | 0 | 0 | 0 | 0 | 0
  Diastolic BP: <40 mmHg, Week 6 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in Height at Week 6
Description: Height was measured in inche without shoes, with the participant stood on a flat surface and with chin parallel to the floor.
Time Frame: Baseline, Week 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Placebo | SPD489 5 mg | SPD489 10 mg | SPD489 20 mg | SPD489 30 mg
Number analyzed (Participants) | 41 | 34 | 32 | 33 | 32
Centimeter | 0.7 (1.21) | 0.7 (1.50) | 0.7 (1.08) | 1.0 (1.29) | 0.5 (1.20)

7. Secondary Outcome: Change From Baseline in Body Weight at Week 6
Description: Body weight was measured in percentile without shoes. Body weight percentile was normalized by sex and age using the Centers for Disease Control and Prevention (CDC) growth charts. Body weight percentiles were categorized as lesser than (<) 5th, 5th to < 95th, and greater than or equal to (>=) 95th percentiles. Change from baseline in body weight at Week 6 was reported.
Time Frame: Baseline, Week 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Weight percentile
Arm/Group | Placebo | SPD489 5 mg | SPD489 10 mg | SPD489 20 mg | SPD489 30 mg
Number analyzed (Participants) | 41 | 34 | 32 | 33 | 32
Weight percentile | -1.1 (5.94) | -1.0 (8.00) | -2.8 (6.37) | -4.8 (9.59) | -5.8 (8.05)

8. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Week 6
Description: BMI was derived from height and weight. BMI percentile was normalized by sex and age using the CDC growth charts. BMI percentiles were categorized as: Underweight (BMI < 5th percentile); Healthy weight (BMI 5th percentile up to < 85th percentile); Overweight (BMI 85th percentile < 95th percentile); Obese (BMI >= 95th percentile). Change from baseline in body mass index at Week 6 was reported.
Time Frame: Baseline, Week 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: BMI percentile
Arm/Group | Placebo | SPD489 5 mg | SPD489 10 mg | SPD489 20 mg | SPD489 30 mg
Number analyzed (Participants) | 41 | 34 | 32 | 33 | 32
BMI percentile | -1.6 (11.17) | -0.9 (14.06) | -5.1 (10.49) | -6.7 (14.28) | -7.4 (11.91)

9. Secondary Outcome: Number of Participants With Potentially Clinically Significant Changes in Clinical Laboratory Values
Description: Clinical laboratory evaluations included biochemistry and endocrinology, hematology, and urinalysis. Number of participants with potentially clinically significant changes in clinical laboratory values were reported. ULN in measure data represents upper limit of normal, mcmol/L represents to Micromoles Per Litre, > = represents greater than or equal to.
Time Frame: Week 6
Population: Safety analysis set consisted of all randomized set who had taken at least 1 dose of investigational product. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure and at the specific categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SPD489 5 mg | SPD489 10 mg | SPD489 20 mg | SPD489 30 mg
Number analyzed (Participants) | 38 | 33 | 31 | 30 | 28
Participants
  Eosinophils/Leukocytes: Greater than (>)10%: number analyzed (Participants) | 37 | 30 | 31 | 27 | 28
  Eosinophils/Leukocytes: Greater than (>)10% | 1 | 0 | 2 | 5 | 0
  Lymphocytes/Leukocytes: Greater than (>) 70%: number analyzed (Participants) | 37 | 30 | 31 | 27 | 28
  Lymphocytes/Leukocytes: Greater than (>) 70% | 1 | 0 | 0 | 0 | 0
  Neutrophils/Leukocytes: Less than (<) 30%: number analyzed (Participants) | 37 | 30 | 31 | 27 | 28
  Neutrophils/Leukocytes: Less than (<) 30% | 6 | 2 | 1 | 3 | 1
  Platelets: >600x10^9/Litre (L): number analyzed (Participants) | 36 | 30 | 30 | 25 | 27
  Platelets: >600x10^9/Litre (L) | 0 | 0 | 0 | 0 | 1
  Alanine aminotransferase: >= 3x ULN: number analyzed (Participants) | 38 | 33 | 31 | 26 | 28
  Alanine aminotransferase: >= 3x ULN | 1 | 0 | 0 | 0 | 0
  Aspartate aminotransferase: >=3x ULN: number analyzed (Participants) | 38 | 33 | 31 | 26 | 28
  Aspartate aminotransferase: >=3x ULN | 1 | 0 | 0 | 0 | 0
  Creatinine: >176.8 mcmol/L or >1.5x ULN: number analyzed (Participants) | 38 | 33 | 31 | 26 | 28
  Creatinine: >176.8 mcmol/L or >1.5x ULN | 0 | 0 | 0 | 1 | 0
  Glucose: <3.05 Millimole per liter (mmol/L): number analyzed (Participants) | 38 | 33 | 31 | 26 | 28
  Glucose: <3.05 Millimole per liter (mmol/L) | 1 | 1 | 0 | 0 | 0
  Glucose: >8.88 Millimole per liter (mmol/L): number analyzed (Participants) | 38 | 33 | 31 | 26 | 28
  Glucose: >8.88 Millimole per liter (mmol/L) | 0 | 0 | 1 | 0 | 0
  Potassium: >5.5 Millimole per liter (mmol/L): number analyzed (Participants) | 38 | 33 | 31 | 26 | 28
  Potassium: >5.5 Millimole per liter (mmol/L) | 1 | 0 | 0 | 0 | 0
  Ketones: Positive value (excluding trace): number analyzed (Participants) | 37 | 33 | 31 | 30 | 27
  Ketones: Positive value (excluding trace) | 1 | 0 | 2 | 3 | 3
  Occult blood: Positive value (excluding trace): number analyzed (Participants) | 37 | 33 | 31 | 30 | 27
  Occult blood: Positive value (excluding trace) | 1 | 0 | 1 | 1 | 3
  Protein: Positive value (excluding trace): number analyzed (Participants) | 37 | 33 | 31 | 30 | 27
  Protein: Positive value (excluding trace) | 7 | 1 | 3 | 4 | 5

10. Secondary Outcome: Number of Participants With Potentially Clinically Significant Changes in Electrocardiogram (ECG) Parameters
Description: Number of participants with potentially clinically significant changes in ECG parameters were reported. QTcF interval represents QT Fridericia's Correction Formula interval, QTcB interval represents QTc corrected by Bazett's in measure data.
Time Frame: Week 6
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SPD489 5 mg | SPD489 10 mg | SPD489 20 mg | SPD489 30 mg
Number analyzed (Participants) | 41 | 34 | 31 | 32 | 32
Participants
  Heart Rate (< 55 Beats per minute) | 0 | 0 | 0 | 0 | 0
  Heart Rate (> 130 Beats per minute) | 0 | 0 | 0 | 0 | 0
  QRS Interval (> = 90 millisecond [msec]) | 1 | 1 | 0 | 1 | 2
  QT Interval (> = 440 msec) | 0 | 0 | 0 | 0 | 0
  QTcB Interval (> =440 msec and <480 msec) | 1 | 1 | 2 | 3 | 2
  QTcB Interval (>=480 msec and <500 msec) | 0 | 0 | 0 | 0 | 0
  QTcB Interval (>=500 msec) | 0 | 0 | 0 | 0 | 0
  QTcF Interval (> =440 msec and <480 msec) | 0 | 0 | 0 | 0 | 0
  QTcF Interval (>=480 msec and <500 msec) | 0 | 0 | 0 | 0 | 0
  QTcF Interval (>=500 msec) | 0 | 0 | 0 | 0 | 0
  ECG Abnormality - Rhythm: number analyzed (Participants) | 4 | 4 | 3 | 3 | 4
  ECG Abnormality - Rhythm | 0 | 1 | 0 | 0 | 0

11. Secondary Outcome: Children's Sleep Habits Questionnaire (CSHQ) at Week 6
Description: Children's Sleep Habits Questionnaire was a tool designed to screen the most common sleep problems in children, and consisted of 33 items for scoring. The instrument evaluated the child's sleep based on behavior within 8 different subscales: bedtime resistance, sleep-onset delay, sleep duration, sleep anxiety, night walkings, parasomnias, sleep-disordered breathing, and daytime sleepiness. Each item receives a score from 1 (problem occurs rarely) to 3 (problem usually occurs); therefore, a higher score is the worse outcome. Scale ranges are as follows: bedtime resistance: 6 to 18, sleep onset delay: 1 to 3, sleep duration: 3 to 9, sleep anxiety: 4 to 12, night walkings: 3 to 9, parasomnias: 7 to 21, sleep-disordered breathing: 3 to 9, daytime sleepiness: 8 to 24, and total disturbance (items from all scales): 33 to 99.
Time Frame: Week 6
Population: Safety analysis set consisted of all randomized set who had taken at least 1 dose of investigational product. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure at the specific categories.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | SPD489 5 mg | SPD489 10 mg | SPD489 20 mg | SPD489 30 mg
Number analyzed (Participants) | 45 | 39 | 35 | 34 | 38
Score on scale
  Bedtime resistance: Week 6: number analyzed (Participants) | 41 | 34 | 32 | 33 | 32
  Bedtime resistance: Week 6 | 9.7 (3.22) | 9.4 (3.30) | 10.3 (3.36) | 10.2 (3.60) | 10.3 (3.30)
  Sleep-onset delay: Week 6: number analyzed (Participants) | 41 | 34 | 32 | 33 | 32
  Sleep-onset delay: Week 6 | 1.7 (0.74) | 1.7 (0.80) | 1.8 (0.75) | 1.8 (0.75) | 1.8 (0.76)
  Sleep duration: Week 6: number analyzed (Participants) | 41 | 34 | 32 | 33 | 32
  Sleep duration: Week 6 | 3.9 (1.20) | 3.9 (1.20) | 3.9 (1.35) | 4.1 (1.70) | 4.1 (1.62)
  Sleep anxiety: Week 6: number analyzed (Participants) | 41 | 34 | 32 | 31 | 31
  Sleep anxiety: Week 6 | 5.7 (2.37) | 5.8 (2.17) | 6.5 (2.36) | 6.5 (2.75) | 6.4 (2.37)
  Night wakings: Week 6: number analyzed (Participants) | 40 | 34 | 32 | 33 | 32
  Night wakings: Week 6 | 4.7 (1.78) | 4.2 (1.23) | 4.6 (1.58) | 4.3 (1.36) | 4.1 (1.39)
  Parasomnias: Week 6: number analyzed (Participants) | 41 | 34 | 32 | 33 | 32
  Parasomnias: Week 6 | 8.6 (1.97) | 8.9 (1.70) | 8.8 (1.50) | 8.2 (1.54) | 8.4 (1.34)
  Sleep-disordered breathing: Week 6: number analyzed (Participants) | 41 | 34 | 32 | 33 | 32
  Sleep-disordered breathing: Week 6 | 3.5 (1.00) | 3.6 (1.02) | 3.3 (0.68) | 3.4 (0.70) | 3.5 (0.95)
  Daytime sleepiness: Week 6: number analyzed (Participants) | 41 | 34 | 32 | 33 | 32
  Daytime sleepiness: Week 6 | 10.9 (3.58) | 10.9 (3.33) | 10.3 (3.33) | 9.8 (3.57) | 12.4 (4.46)

12. Secondary Outcome: Number of Participants With a Positive Response Using Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS was semi-structured interview that captured the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The interview included definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behavior occurred. The C-SSRS contained 2 required items pertaining to suicidal ideation, 4 required items pertaining to suicidal behavior, and 1 required item pertaining to non-suicidal but self-injurious behavior. In situations where there was a positive response to the screening questions, there were 8 additional suicidal ideation items and 4 additional suicidal behavior items which were completed. Thus, there was a maximum of 19 items to be completed. Here number of participants responded as yes to suicidal ideation or behaviour were reported.
Time Frame: Up to Week 6
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Placebo | SPD489 5 mg | SPD489 10 mg | SPD489 20 mg | SPD489 30 mg
Number analyzed (Participants) | 45 | 39 | 34 | 34 | 38
Participants | 0 | 1 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: From start of the study drug administration up to follow up (Week 7)
Groups:
- SPD489 5 mg: Participants received SPD489 capsule orally at a dose of 5 milligram (mg) once daily for 6 weeks.
- SPD489 10 mg: Participants received SPD489 capsule orally at a dose of 10 mg once daily for 6 weeks.
- SPD489 20 mg: Participants received SPD489 capsule orally at a dose of 20 mg once daily for 6 weeks.
- SPD489 30 mg: Participants received SPD489 capsule orally at a dose of 30 mg once daily for 6 weeks.
Arm/Group | Placebo | SPD489 5 mg | SPD489 10 mg | SPD489 20 mg | SPD489 30 mg
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/39 | 0/35 | 0/34 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/39 | 0/35 | 0/34 | 0/38
Other Adverse Events (participants affected / at risk) | 4/45 | 8/39 | 11/35 | 14/34 | 18/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=45) | SPD489 5 mg (N=39) | SPD489 10 mg (N=35) | SPD489 20 mg (N=34) | SPD489 30 mg (N=38)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 3 (3) | 6 (6) | 8 (8)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Affect lability (Psychiatric disorders) | 0 (0) | 2 (2) | 3 (4) | 1 (1) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Irritability (Psychiatric disorders) | 0 (0) | 3 (3) | 4 (4) | 3 (3) | 4 (4)
Middle insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT03260205/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/05/NCT03260205/SAP_001.pdf